CLINICAL TRIAL: NCT01863914
Title: Effect of Rosuvastatin in the Mobilization of Endothelial Progenitor Cells and Graft Vascular Function Following Creation of Arteriovenous Fistula in Diabetic Patients With Chronic Renal Failure
Brief Title: Vascular Protective Effect of Rosuvastatin in Arteriovenous Fistula
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Lam Chen Fuh, Associate Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 101-2314-B-006-045
Record Dates: First submitted 2013-02-14; First posted 2013-05-29 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: End-stage Kidney Disease; Diabetes Mellitus; Arteriovenous Fistula
Keywords: ESRD; Diabetes mellitus; Endothelial progenitor cells; Hemodialysis; rosuvastatin
MeSH Terms: conditions — Kidney Failure, Chronic; Diabetes Mellitus; Arteriovenous Fistula | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablet contains only inactive ingredient. The placebo tablets will be taken once daily for 4 weeks (1 week before operation and 3 weeks after creation of AV fistula)
  Interventions: Drug: Rosuvastatin
- Rosuvastatin (Active Comparator): Rosuvastatin (CrestorÒ, Astrazeneca) 5mg once daily for 4 weeks (1 week before operation and 3 weeks after creation of AV fistula)
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Arteriovenous fistula surgery was performed after 1-week treatment with placebo or Rosuvastatin (randomized, double blind). The intervention drug treatment continues for 3 more weeks after creation of AV fistula.
  Other Names: Crestor

SUMMARY:
Background Arteriovenous (AV) fistula is the most common vascular access for long-term hemodialysis in the end-stage renal disease (ESRD) patients. About 25% of these patients are diabetes mellitus. However, the effects of hyperglycemia on the vascular function of arteriovenous fistula are still remained unclear. Studies have shown that blood flow in the AV fistula is significantly reduced in patients with diabetes mellitus. Diabetic patients also require a longer period of time for the maturation of AV fistula, and have slightly higher complication rate than non-diabetic patients. Statins have been widely shown to mediate several important pleiotropic effects in the improvement of vascular endothelial dysfunction, attenuation of inflammatory responses, stabilization of atherosclerotic plaques, inhibition of vascular smooth muscle proliferation, and modulation of procoagulant activity and platelet function.Our experimental studies in diabetic animals demonstrate that administration of a water-soluble statin rosuvastatin significantly improves the fistula flow, vascular function and luminal dilatation of AV fistula in diabetic rats by suppression of vascular oxidative stress and inflammatory load.

Study hypothesis The central hypothesis of this research project is rosuvastatin mediates pleiotropic protective effect on vascular endothelial function and suppresses the regional pro-inflammatory reaction in the vasculature, therefore administration of rosuvastatin during the perioperative period of creation of native AV fistulas in diabetic patients with ESRD may potentiate the vascular function and reduce the primary failure rate of AV fistulae.

DETAILED DESCRIPTION:
Background In Taiwan, diabetic nephropathy is the second most common cause of end-stage renal disease (ESRD), but diabetic patients engender 12% more expense for care of dialysis than non-diabetic patients. ESRD patients with diabetes are also more frequently hospitalized due to problems such as failure of vascular access. Hemodialysis necessitates the placement of an arteriovenous (AV) fistula, which involves a direct anastomosis of the radial/brachial artery and cephalic vein. In the United States, procedures for creating the AV fistula and treatment of the related complication account for over 20% of hospitalizations of dialysis patients and cost about US$100 million annually. Two major hurdles in establishing a useable and patent AV fistula for dialysis are primary failure (failure of fistula to mature adequately for dialysis) and long-term survival of the vascular access. The reported primary failure rate varies from 20 to 50%. It has been shown that reduction of blood flow (>15% drop of flow over time) is the most critical factor for premature failure of AV fistula. Although blood flow in the venous site of AV fistula is also determined by the surrounding draining veins, blood pumped from the arterial site is the most important factor in maintaining sufficient fistula blood flow. However, very limited of studies have reported the effect of arterial blood flow on the function and patency of AV fistula. More evidences have shown that progressive failure of AV fistula after long-term use is due to the development of thrombosis (~80%) and stenosis (~20%). The mechanisms that underlie the failure of AV fistula are still poorly understood and there are very few, if any, specific therapeutic approaches that can increase the lifespan of these fistulas. Therefore, there is the critical need for experimental studies that seek to understand the basic mechanisms of primary failure and progressive failure of the AV fistula in diabetes mellitus.

Creation of an AV fistula is the most common vascular access for ESRD patients, who require long-term hemodialysis. In Taiwan, about 25% of these patients have underlying diabetes mellitus. However, the effects of hyperglycemia on the vascular function of arteriovenous fistula are still remained unclear. Studies have shown that blood flow in the AV fistula is significantly reduced in patients with diabetes mellitus. Diabetic patients also require a significantly longer period of time (2 more months) for the maturation of AV fistula, and have slightly higher complication rate than non-diabetic patients. Diabetes mellitus has been shown as an independent risk factor of reduced blood flow in the native vessel arteriovenous fistula. Compared with patients without diabetes access blood flow was significantly lower in patients with diabetes mellitus (788±580 vs 1054±681 ml/min, P = 0.002). Patients with diabetes mellitus required a longer time until first use of their AV fistula than did patients without diabetes (4.4±2.9 vs 2.9±1.6 months, respectively, P= 0.02). AV access-related complications and need of re-intervention were higher in these patients. Most recently, Previous study identified that risk for reduced primary patency of AV fistula was increased by diabetes (Hazard Ratio, 1.54; 95% Confidence Interval, 1.14-2.07). Presence of diabetes is also a strong independent predictive factor for reduced initial intra-access blood flow within 6 months after creation of AV fistula (OR 3.5, P = 0.001). However, there is currently very limited effective therapeutic strategy in the prevention of loss of primary patency and improvement of life expectancy of AV access in patients with diabetes.

3-Hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase inhibitors (statins) are one of the most commonly prescribed agents in controlling hyperlipidemia. Apart from their serum lipid-lowering properties, statins have been widely shown to mediate several important pleiotropic effects, such as improvement of vascular endothelial dysfunction, attenuation of inflammatory responses, stabilization of atherosclerotic plaques, inhibition of vascular smooth muscle proliferation, and modulation of procoagulant activity and platelet function. Among these pleiotropic effects, the protective effects on vascular endothelial function have mostly been highlighted. In clinical settings, statins improve cardiovascular outcomes of patients with atherosclerosis even in the population of normal plasma cholesterol level. The improvement in cardiovascular outcomes is well correlated with improved endothelial function by upregulation of endothelial nitric oxide synthase (eNOS) expression and nitric oxide (NO) bioavailability following treatment with statins. At subcellular levels, statins stabilize the eNOS messenger ribonucleic acid (mRNA), enhance eNOS enzymatic activity via phosphatidyl inositide (PI)3 kinase signaling pathway, reduce inflammatory responses in the vasculature, inhibit Rho isoprenylation and suppress oxidized- LDL-induced endothelin-1 expression. Statins have also been characterized to enhance re-endothelialization of damaged vascular endothelium by stimulating pre-existing endothelial cells and by mobilizing bone marrow-derived endothelial progenitor cells (EPCs). Collectively, stains restore vascular endothelial function and mediate vascular protective effects that are independent from their lipid-lowering effects. Although the beneficial pleiotropisms by statins are well documented in a variety of endothelial dysfunctional disorders, their potential therapeutic effects in maintaining a healthy, usable AV fistula in subjects with diabetes mellitus have been previously demonstrated.

According to the knowledge of applicant, there was no published randomized control clinical study prospectively investigated the vascular protective effect of statins on the establishment of AV fistula in patients with chronic kidney disease (CKD) or ESRD. A long-term (up to 987 days) case-control study suggested that patients receiving statin therapy were associated with significantly higher overall primary patency rate of AV fistula after 1 year (81.7 vs 66 %) and after 2 years (71.5 vs 39.1%).

During the past national science council (NSC)-funded years 2009-2011, the applicant undertook experimental study in rats with streptozotocin-induced diabetes, in which an AV fistula was created in each control and diabetic animals. The diabetic rats received either placebo or rosuvastatin (10 mg/kg/d) in chow for a period 18 days (3 days before creation of AV fistula and 14 after operation). Circulating cluster of differentiation (CD)133+/vascular endothelial growth factor receptor (KDR)+ EPCs were determined 2 weeks after creation of AV fistula using flow cytometry. Vascular function of AV fistula was assessed by isometric force testing. The expression of pro-inflammatory genes (iNOS and NADPH oxidase) and generation of superoxide anions in the fistula were examined. The results showed that number of EPCs was reduced in diabetic rats, and rosuvastatin significantly increased numbers of circulating EPC. Reduced blood flow and impaired endothelium-dependent relaxation in the AV fistula of animals with diabetes was significantly potentiated following treatment with rosuvastatin. Rosuvastatin also attenuated the expression of iNOS and NADPH oxidase, and generation of superoxide anions in the fistula tissues isolated from diabetic rats. These findings provide the first and very important evidence demonstrating that rosuvastatin improves blood flow and endothelial function of AV fistula in subjects with diabetes mellitus by attenuating the activity of pro-inflammatory genes and generation of superoxide anions in the remodeled vasculature. Based on these fascinating and encouraging findings, the applicant proposes to undertake clinical study in translating these experimental results to diabetic patients with CKD, who are scheduled to creation of AV fistula for further hemodialysis.

Central Hypothesis and Specific Aims

The central hypothesis of this research project is rosuvastatin mediates pleiotropic protective effect on vascular endothelial function and suppresses the regional pro-inflammatory reaction in the vasculature, therefore administration of rosuvastatin during the perioperative period of creation of native AV fistulas in diabetic patients with ESRD may potentiate the vascular function and reduce the primary failure rate of AV fistulae. Here, the applicant proposes to undertake a three-year research project investigating the therapeutic potential of rosuvastatin in the establishment of AV fistula in patients with diabetes mellitus. The applicant opts to test the proposed effect of rosuvastatin in diabetic patients. The long-term aim of this project is to develop a clinical feasible, endothelium-targeted therapeutic strategy for a durable AV fistula in human subjects necessitates hemodialysis. To achieve these research goals the applicant proposes studies with following specific aims:

1. Administration of rosuvastatin protects the endothelial function in the AV fistula and restores the blood flow rate in the shunt of diabetic patients with ESRD, thereby improves the primary patent rate and early maturation of these fistulas.
2. Administration of rosuvastatin improves the vascular function of AV fistulas in diabetic patients with ESRD, therefore reduces the overall shunt-related complication rate and the requirement for surgical re-interventions.
3. Administration of rosuvastatin is associated with reduction of the systemic pro-inflammatory response and oxidative stress (levels of proinflammatory cytokines and other mediators in the circulation) in diabetic patients with ESRD. On the other hand, administration of rosuvastatin may mobilize the bone marrow-derived EPCs into systemic circulation, and the number of these circulating endothelial progenitors may provide prognostic value to the outcomes of AV fistula.
4. Administration of rosuvastatin reduces the overall perioperative cardiovascular and other morbidities in diabetic patients with ESRD.
5. Administration of rosuvastatin does not increase the incidence of statin-related complications (such as myopathy, abnormal liver function and neurologic deficit) in diabetic patients with ESRD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diabetes mellitus (postprandial blood sugar >140 mg/dl)
2. Patients with end-stage kidney disease and is proposed to undertake chronic hemodialysis
3. Patients of age 18-65 years
4. The fistula is constructed in the forearm (radiocephalic fistula).

Exclusion Criteria:

1. Preoperative blood sugar level >250 mg/dl or most recent HbA1c >10%
2. Recent treatment with statins within 2 weeks before evaluation for clinical trial
3. Advanced liver disease
4. Chronic alcoholism
5. Congestive heart failure
6. Coronary disease which require permanent statin therapy
7. Malignancy or hematologic disorder
8. Pregnancy or breastfeeding
9. Past history of creation of AV fistula
10. Scheduled for general anesthesia
11. Emergent operation
12. peripheral arterial occlusion disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Primary patent rate of AV fistula | 6 months after operation
  The definition of primary patency of an AV fistula is defined as successful cannulation of the fistula for first hemodialysis treatment (first dialysis session)(reference: BioMed Central Nephrology 2013;14:79). Administration of rosuvastatin protects the endothelial function in the AV fistula and restores the blood flow rate in the shunt of diabetic patients with ESRD, thereby improves the primary patent rate and early maturation of these fistulas

SECONDARY OUTCOMES:
Composite outcome measurement of the overall shunt-related complication rate | 6 months after operation
  The most commonly shunt-related complications are formation of aneurysms, failure of shunt to mature, and development of thrombosis in AV fistula (Ann Vasc Surg 2012;26:680). The occurrence of shunt-related complications usually require surgical reintervention. Administration of rosuvastatin improves the vascular function of AV fistulas in diabetic patients with ESRD, therefore reduces the overall shunt-related complication rate and the requirement for surgical re-interventions.

OTHER OUTCOMES:
Composite outcome measurement of systemic pro-inflammatory response | 6 months after operation
  Systemic proinflammatory response is determined by measuring blood concentrations of monocyte chemo-attractant protein (MCP)-1, interleukin (IL)-1 beta, IL-6 and tumor necrosis factor (TNF)-alpha, and the numbers of circulating endothelial progenitor cells (EPCs). Administration of rosuvastatin is associated with reduction of the systemic pro-inflammatory response and oxidative stress (levels of proinflammatory cytokines and other mediators in the circulation) in diabetic patients with ESRD. On the other hand, administration of rosuvastatin may mobilize the bone marrow-derived EPCs into systemic circulation, and the number of these circulating endothelial progenitors may provide prognostic value to the outcomes of AV fistula.

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Neng Roan, MD, PhD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The Ethical committee in National Cheng Kung University Hospital approved major modification of a reduction of case collection from 80 to 60 cases on 2018-8-9. The study had recruited a total of 60 cases in the trial before 2018-12-31. The results were under analysis by the statistician. Moreover, exposure of the treatment group and placebo group were not performed until after completion of data analysis by the statistician in early February. The results might be revealed as appropriate in the website.

REFERENCES:
- [Background] Roan JN, Fang SY, Chang SW, Hsu CH, Huang CC, Chiou MH, Tsai YC, Lam CF. Rosuvastatin improves vascular function of arteriovenous fistula in a diabetic rat model. J Vasc Surg. 2012 Nov;56(5):1381-9.e1. doi: 10.1016/j.jvs.2012.03.243. Epub 2012 Jun 22. PMID 22727844
- [Background] Fang SY, Roan JN, Lin Y, Hsu CH, Chang SW, Huang CC, Tsai YC, Lam CF. Rosuvastatin suppresses the oxidative response in the venous limb of an arteriovenous fistula and enhances the fistula blood flow in diabetic rats. J Vasc Res. 2014;51(2):81-9. doi: 10.1159/000357619. Epub 2014 Jan 15. PMID 24434545